CLINICAL TRIAL: NCT05774249
Title: The Value of Adding Pecto-intercostal Fascial Plane Block on the Postoperative Analgesia and Recovery Profile After Off-Pump Coronary Artery Bypass Surgery
Brief Title: Pecto-intercostal Fascial Plane Block for Postoperative Analgesia and Recovery Profile After Off-Pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R34/2023
Record Dates: First submitted 2023-03-04; First posted 2023-03-17 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided pectointercostal fascial plane block group (Active Comparator): using 20 mL of 0.25% bupivacaine with adrenaline 1:400,000
  Interventions: Procedure: Ultrasound guided pecto-intercostal Fascial Plane Block using bupivacaine
- control group (Placebo Comparator): using 20 mL of normal saline 0.9%
  Interventions: Procedure: Ultrasound guided pecto-intercostal Fascial Plane Block using normal saline

INTERVENTIONS:
Procedure: Ultrasound guided pecto-intercostal Fascial Plane Block using bupivacaine — while Patients in supine decubitus position,parasternal area will be scanned using high frequency ultrasound linear probe .After identification of ribs with intercostal spaces in between ;the fourth intercostal space will be approached via 10 cm block needle targeting the plane between pectoralis major and external intercostal muscle under ultrasound guidance after which 20 mL of 0.25% bupivacaine with adrenaline 1:400,000 will be administered in increments bilaterally.
  Arms: Ultrasound guided pectointercostal fascial plane block group
Procedure: Ultrasound guided pecto-intercostal Fascial Plane Block using normal saline — Sham Block will be done while Patients in supine decubitus position,parasternal area will be scanned using high frequency ultrasound linear probe .After identification of ribs with intercostal spaces in between ;the fourth intercostal space will be approached via 10 cm block needle targeting the plane between pectoralis major and external intercostal muscle under ultrasound guidance after which 20 mL of normal saline 0.9 % will be administered bilaterally.
  Arms: control group

SUMMARY:
Moderate to severe postoperative pain is usually encountered after cardiac surgery.Improper postoperative pain control could have multiple hemodynamic hazards in addition to prolonged postoperative ventilatory support and intensive care unit stay .The safety and efficacy of ultrasound guided chest wall plane blocks has been described for postoperative analgesia after cardiac surgeries.

Study objective: to investigate the effect of adding of pecto-intercostal fascial plane block on the postoperative pain control, perioperative analgesic consumptions and the time for ventilation weaning and intensive care unit discharge in patients who will undergo off-pump Coronary artery bypass surgeries.

Methods: This study patients will be randomly assigned to 2 Groups to receive preoperative ultrasound-guided pecto-intercostal fascial plane block with either 20 mL of 0.25% bupivacaine with adrenaline 1:400,000 or saline bilaterally.

DETAILED DESCRIPTION:
After preoperative patients' anesthesia assessment; the study patients (20 in each group) will receive general anesthesia under invasive monitoring of hemodynamics, and oxygen saturation. After anesthesia induction; cannulation of jugular vein and insertion of transoesophageal echocardiography and temperature probe will be done. In block group : while Patients in supine decubitus position,parasternal area will be scanned using high frequency ultrasound linear probe .After identification of ribs with intercostal spaces in between ;the fourth intercostal space will be approached via 10 cm block needle targeting the plane between pectoralis major and external intercostal muscle under ultrasound guidance after which 20 mL of 0.25% bupivacaine with adrenaline 1:400,000 will be administered in increments bilaterally. In control group:Sham Block will be done using 20 mL of normal saline 0.9% bilaterally .

Anesthesia will be maintained with sevoflurane inhalational anesthesia and incremental cisatracurium and fentanyl for intraoperative muscle relaxation and analgesia respectively. Intraoperative anticoagulation will be carried out before revascularization using intravenous heparin titrated according to activated clotting time ,which will be reversed after end of surgery using protamine sulfate.

At the end of surgery patients will be sent to post cardiac surgery intensive care unit . Postoperative analgesia in the form of intravenous paracetamol one gram will be administered on intensive care unit admission then fentanyl based patient controlled analgesia will be started . IV tramadol 1mg/kg as second rescue analgesia will be given if visual analogue scores are still ≥ 4.

ELIGIBILITY:
Inclusion Criteria:

* NYHA ( New york heart association ) class I- III

Exclusion Criteria:

* Parents' refusal to study participation.
* Patients with poor coronary vessels targets.
* Patients with poor cardiac systolic function or preoperative hemodynamic unstability
* Redo coronary artery bypass surgery
* Intraoperative complication need conversion to on pump surgery
* Postoperative exploration for bleeding or poor coronary revascularization
* Advanced COPD(chronic obstructive pulmonary disease) patients.
* Myopathies and myasthenic patients
* Allergy to study medications

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
visual analogue score | immediately after extubation
  0 (no pain) and 10 (worst possible pain)
visual analogue score | 1 st hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 2 nd hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 4 th hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 8 th hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 12 th hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 18 th hour after extubation
  0 (no pain) and 100 (worst possible pain)
visual analogue score | 24 th hour after extubation
  0 (no pain) and 100 (worst possible pain)

SECONDARY OUTCOMES:
Total intraoperative opioid consumption | during the operation
Total postoperative opioid consumption | 24 hour after operation
Number of patients need postoperative rescue tramadol | 24 hours after extubation
Time to patient extubation | at the end of surgery
time for ICU discharge | 72 hours after surgery
postoperative complication | 72 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt